CLINICAL TRIAL: NCT03388320
Title: Using Addiction Comprehensive Health Enhancement Support System (ACHESS) in an Alcoholic Liver Disease Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Nicole T Shen, Principal Investigator, New York Presbyterian Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1704018122
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Liver Diseases, Alcoholic
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving A-CHESS (Experimental): Participants will be provided access to the smartphone application A-CHESS (intervention) that will be downloaded to their phone.
  Interventions: Device: A-CHESS

INTERVENTIONS:
Device: A-CHESS — Use of smartphone application: Addiction Comprehensive Health Enhancement Support System (A-CHESS)

SUMMARY:
This is a pilot study examining whether an evidence-based recovery support smartphone application, the Addiction Comprehensive Health Enhancement Support System (A-CHESS), can decrease alcohol recidivism in a previously unstudied group of patients with alcoholic liver disease (ALD).

DETAILED DESCRIPTION:
A-CHESS is a smartphone application developed by the University of Wisconsin-Madison based on self-determination theory, with a previous randomized clinical trial showing that use of the app resulted in significantly fewer risky drinking days in patients leaving treatment for alcohol-use disorders. The application is downloaded to the participant's smartphone, and provides ongoing access to peer support and educational materials, monitoring of the risk of relapse, and delivery of reminders and encouragements to the patient. The application also has a survey platform to assess and reassess the participants' most recent alcohol consumption, quality of life, and experience using the application. We anticipate that use of the A-CHESS app will result in decreased drinking and improved abstinence, identifying a potential intervention to offer patients with ALD to improve their mortality, liver disease, and likelihood of liver transplant candidacy status.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholic liver disease
* Followed or seen at New York Presbyterian Hospital / Weill Cornell Medical Center
* English speaking
* Access to a smartphone

Exclusion Criteria:

* Unable to consent
* Primary language other than English
* No access to a smartphone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Rates of recidivism | 6 months
  Rates of recidivism in this population using A-CHESS will be compared to historical control rates

SECONDARY OUTCOMES:
Use of A-CHESS | 6 months
  The association between the extent to which patients use the A-CHESS application and their recidivism; to compare use of the A-CHESS app among subjects who drink and remain abstinent.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brown, MD, MPH, Principal Investigator — Weill Cornell Medical College/NYPH
Locations (1):
- New York Presbyterian Hospital - Weill Cornell Medicine and Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No